CLINICAL TRIAL: NCT00001116
Title: Effect of Recombinant Human Soluble Tumor Necrosis Factor Receptor (TNFR:Fc) on Interleukin-6 (IL-6), Tumor Necrosis Factor-Alpha (TNF-alpha) and Markers of Immune Activation in HIV-Infected Subjects
Brief Title: A Study to Evaluate the Ability of TNFR:Fc to Decrease the Amount of IL-6 (Interleukin-6) and TNF-alpha (Tumor Necrosis Factor) in HIV-Infected Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: ACTG 928; 11498 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Tumor Necrosis Factor; Interleukin-2; Immunity, Cellular; Antiviral Agents; Interleukin-6; Receptors, Tumor Necrosis Factor
MeSH Terms: conditions — HIV Infections

INTERVENTIONS:
Drug: Tumor Necrosis Factor soluble receptor-immunoadhesin complex

SUMMARY:
The purpose of this study is to determine if TNFR:Fc (a molecule that attaches to TNF) can lower the amount of IL-6 in HIV-positive patients. This study will also examine the effect of TNFR:Fc on TNF-alpha. IL-6 and TNF-alpha are 2 substances produced by the immune system that may increase the rate of HIV replication.

IL-6 and TNF-alpha are produced naturally by the body. High levels of TNF-alpha lead to increased IL-6 production and increased HIV replication, therefore helping the virus infect the body. HIV-positive patients who receive IL-2 (interleukin-2, a protein that helps the immune system fight infection) tend to have higher levels of IL-6 and TNF-alpha than patients not receiving IL-2. These increased levels may contribute to some of the flu-like symptoms related to IL-2 administration. TNFR:Fc can neutralize TNF-alpha to decrease the action of TNF-alpha and, in turn, decrease the amount of IL-6 in the body. TNFR:Fc may, therefore, have a role in the treatment of HIV disease or in relieving some of the symptoms related to IL-2 administration.

DETAILED DESCRIPTION:
Both Interleukin-6 (IL-6) and Tumor necrosis factor-alpha (TNF-alpha) are substances naturally produced by the body's immune system. Evidence suggests that TNF-alpha production may be excessive or inappropriate in HIV-infected patients. Elevated TNF-alpha levels can result in increased IL-6 production and possibly increased HIV replication. TNFR:Fc is a modification of a natural substance that binds to TNF-alpha and neutralizes its activity. It is postulated that TNFR:Fc may result in decreased activity of TNF-alpha and lower IL-6 levels. HIV-infected patients who receive Interleukin-2 (IL-2) have been shown to have higher TNF-alpha and IL-6 levels than those who do not receive IL-2. It is thought that these higher levels of TNF-alpha and IL-6 may contribute to some of the flu-like symptoms experienced by patients receiving IL-2. By decreasing the amount of IL-6 in the body and by decreasing the action of TNF-alpha in the body, TNFR:Fc may have a role in the treatment of HIV disease or in alleviating some of the symptoms related to IL-2 administration.

Six patients from each of the 3 treatment arms of ACTG 328 (HAART alone, HAART plus intravenous (IV) rhIL-2, and HAART plus subcutaneous (SC) rhIL-2) who are about to be randomized to Step II of ACTG 328 may participate in this prospective, nested substudy. Patients randomized to the Interleukin-2 (IL-2) arms of ACTG 328 are pretreated with TNFR:Fc (administered by infusion over 30 minutes) at week 16 of ACTG 928 (Course 3, Week 28 of ACTG 328), just prior to initiation of IL-2. Those randomized to the highly active antiretroviral therapy (HAART) only arm of ACTG 328 receive treatment with TNFR:Fc at Week 16 of ACTG 928 (Week 28 of ACTG 328).

ELIGIBILITY:
Inclusion Criteria

You may be eligible for this study if you:

* Are HIV-positive.
* Are enrolled in ACTG 328.
* Agree to practice abstinence or use barrier methods of birth control during the study.
* Are at least 18 years old.

Exclusion Criteria

You will not be eligible for this study if you:

* Have any active opportunistic (HIV-associated) infections.
* Have any medical condition or psychological issue that would interfere with study requirements.
* Are pregnant or breast-feeding.
* Are receiving any experimental drug other than IL-2.
* Are receiving certain other medications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18
Dates: Study Completion 2000-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sha B, Study Chair; Valdez H, Study Chair; Landay A, Study Chair; Lederman M, Study Chair
Locations (3):
- United States (3):
  - Univ. of Hawaii at Manoa, Leahi Hosp., Honolulu, Hawaii
  - NY Univ. HIV/AIDS CRS, New York, New York
  - Case CRS, Cleveland, Ohio

REFERENCES:
- [Background] Lange CG, Valdez H, Medvik K, Asaad R, Lederman MM. CD4+ T-lymphocyte nadir and the effect of highly active antiretroviral therapy on phenotypic and functional immune restoration in HIV-1 infection. Clin Immunol. 2002 Feb;102(2):154-61. doi: 10.1006/clim.2001.5164. PMID 11846457
- [Background] Sha B, Valdez H, Landay A, Gelman R, Namkung A, Agosti J, Bancroft L, Mildvan D, Mitsuyasu R, Pollard R, Ogata-Arakaki D, Kilgo P, Estep S, Fox L, Lederman M. Effect of recombinant human soluble tumor necrosis factor receptor (TNFR, etanercept) on interleukin-6 (IL- 6), TNF-a, and markers of immune activation in HIV-infected subjects receiving interleukin-2 (IL-2). 8th Conf Retro and Opportun Infect. 2001 Feb 4-8 (abstract no 66)
- [Background] Sha BE, Valdez H, Gelman RS, Landay AL, Agosti J, Mitsuyasu R, Pollard RB, Mildvan D, Namkung A, Ogata-Arakaki DM, Fox L, Estep S, Erice A, Kilgo P, Walker RE, Bancroft L, Lederman MM. Effect of etanercept (Enbrel) on interleukin 6, tumor necrosis factor alpha, and markers of immune activation in HIV-infected subjects receiving interleukin 2. AIDS Res Hum Retroviruses. 2002 Jun 10;18(9):661-5. doi: 10.1089/088922202760019365. PMID 12079562